CLINICAL TRIAL: NCT00262431
Title: Efficacy of Early Tracheostomy to Reduce Incidence of Ventilator Acquired Pneumonia (VAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Regione Piemonte (Other)
Responsible Party: Principal Investigator, Marco Ranieri, MD, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1431/28.3
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Respiratory Insufficiency
Keywords: Tracheostomy; Tracheostomy timing; Ventilator associated pneumonia; Mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia, Ventilator-Associated

ARMS (2):
- Early (A) (Active Comparator): Patients of the EARLY group (A) will be submitted to tracheostomy on day 3-5 from oro/nasotracheal intubation.
  Interventions: Procedure: Tracheostomy on day 3-5 in early group and 10-12 in late group
- Late (B) (Active Comparator): Patients of the LATE group (B) will undergo tracheostomy on day 10-12 from oro/nasotracheal intubation.
  Interventions: Procedure: Tracheostomy on day 3-5 in early group and 10-12 in late group

INTERVENTIONS:
Procedure: Tracheostomy on day 3-5 in early group and 10-12 in late group — Upon admission to ICU, acute respiratory failure patients requiring at least 3 days of mechanical ventilation and defined by a SAPS II score between 35 and 65, will be randomly assigned to either arm A or B of the study.

SUMMARY:
The study aims to assess early (one to three days after intubation) tracheostomy effectiveness in terms of reduction in ventilator associated pneumonia (VAP) incidence.

DETAILED DESCRIPTION:
Tracheostomy is an essential and irreplaceable procedure for critically ill patients requiring mechanical ventilatory support and adequate airway control. The therapeutical choice of performing a tracheostomy is supported by a number of clinical benefits, such as less use of drugs for sedation, fewer days of mechanical ventilation and hence shorter Intensive Care Unit (ICU) length of stay, as well as better resource rationalization. Actually there is no agreement on the best timing for tracheostomy. The aim of this study is to verify if an early tracheostomy (one to three days after intubation) increases ventilator associated pneumonia-free days. Secondary endpoints are: increase of ventilator free-days and mortality reduction.

ELIGIBILITY:
Inclusion Criteria:

* Oro/nasotracheal intubation for less than three days
* Simplified Acute Physiology Score (SAPS II) between 35 and 65 upon admission to Intensive Care Unit (ICU)

Exclusion Criteria:

* Oro/nasotracheal intubation > three days
* Age < 18 years
* Previous otolaryngologic or maxillofacial procedures
* Brain injury patients with intracranial pressure > 20 mmHg without pharmacological treatment (or intracranial pressure > 15 mmHg under specific pharmacological treatment) and with cerebral perfusion pressure < 60 mmHg
* Pregnancy
* Ventilator associated pneumonia, hospital acquired pneumonia, community acquired pneumonia diagnosis before randomization
* Infection in the tracheostomic area
* Acute worsening of chronic obstructive pulmonary disease (COPD)
* Pre-existing malignancies in the tracheostomic area
* Immunosuppressed and/or immunodepressed patients:

  * leukocytes < 1000/microliters
  * neutrophils < 500/microliters
  * AIDS
  * long-term steroid treatment (daily dose > 0.5 mg/kg for more than 30 days)
* Patients already enrolled in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2004-06; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Increase of "ventilator associated pneumonia-free days" | Follow-up terminates on day 28 from the date of oro/nasotracheal intubation.

SECONDARY OUTCOMES:
Increase of "ventilator-free days" | Follow-up terminates on day 28 from the date of oro/nasotracheal intubation
Reduction of mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: V. M. Ranieri, MD, Principal Investigator — University of Turin, Italy; V. M. Ranieri, MD, Study Director — University of Turin, Italy
Locations (1):
- University of Turin, Department of Anesthesia and Intensive Care Medicine, Turin, Italy

REFERENCES:
- [Derived] Terragni PP, Antonelli M, Fumagalli R, Faggiano C, Berardino M, Pallavicini FB, Miletto A, Mangione S, Sinardi AU, Pastorelli M, Vivaldi N, Pasetto A, Della Rocca G, Urbino R, Filippini C, Pagano E, Evangelista A, Ciccone G, Mascia L, Ranieri VM. Early vs late tracheotomy for prevention of pneumonia in mechanically ventilated adult ICU patients: a randomized controlled trial. JAMA. 2010 Apr 21;303(15):1483-9. doi: 10.1001/jama.2010.447. PMID 20407057